CLINICAL TRIAL: NCT03907748
Title: HOMESIDE: Home-based Family Caregiver-delivered Music and Reading Interventions for People Living With Dementia: A Randomised Controlled Trial
Brief Title: Home-based Family Caregiver-delivered Music and Reading Interventions for People With Dementia
Acronym: HOMESIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: University of Melbourne (Other); Norwegian Academy of Music (Other); University of Applied Sciences Würzburg-Schweinfurt (Unknown); University School of Physical Education, Krakow, Poland (Other); Alzheimer's Society (Other); Methodist Homes for the Aged (Other); Saffron Hall Trust (Unknown); Cambridgeshire and Peterborough NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U4-10366; ACTRN12618001799246p (Registry Identifier: Austrailian New Zealand Clinical Trials Registry); 462 (Other Grant/Funding Number: Alzheimer's Society)
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-02

CONDITIONS: Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Dementia, Mixed; Dementia Alzheimers; Behavioural and Psychiatric Symptoms of Dementia; Depression; Quality of Life
Keywords: music therapy; music interventions; home-based interventions; Reading; dementia; care giver
MeSH Terms: conditions — Dementia; Dementia, Vascular; Lewy Body Disease; Mixed Dementias; Alzheimer Disease; Depression

STUDY DESIGN:
Intervention Model Description: Participants (people with dementia and their cohabiting family caregivers) will be allocated to either (1) the music intervention group, (2) the reading intervention group or (3) the standard care group.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be collected by researchers who are not aware of the whether the participants' are allocated to the music, reading or standard care groups. The participants will be reminded not to reveal the group they are in to the person collecting the data. The participants themselves cannot be blinded due to the active nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Intervention (Experimental): The music intervention will be provided to participant dyads (people with dementia and their cohabiting family caregivers) allocated to the first intervention. Caregivers will be trained to use the music intervention in three 2-hour training sessions with an intervention trainer (a music therapist). Training will take place at the dyad's home. The caregiver will then be asked to deliver the music intervention to the person with dementia at least 5x per week for 30 minutes.
  Interventions: Other: Music Intervention
- Reading Intervention (Active Comparator): The reading intervention will be provided to participant dyads (people with dementia and their cohabiting caregivers) allocated to the second intervention. Caregivers will be trained to use the reading intervention in three 2-hour training sessions with an intervention trainer. Training will take place at the dyad's home. The caregiver will then be asked to deliver the reading intervention to the person with dementia at least 5x per week for 30 minutes.
  Interventions: Other: Reading Intervention
- Standard Care (No Intervention): Participant dyads (people with dementia and their cohabiting caregivers) allocated to the standard care group will not receive any training or be asked to deliver an intervention.

INTERVENTIONS:
Other: Music Intervention — After training, caregivers will deliver the music intervention to the person with dementia whom they care for. The music intervention will include: a) singing familiar/preferred music followed by discussions facilitated by the caregiver about any associated meanings or memories; b) movement to music (e.g. upper body and arms imitating familiar dance movements to music); c) instrument playing; and d) listening to familiar/preferred relaxing or enlivening music (dependent upon symptoms present in the moment). These methods are known to assist in emotion regulation and increase cognitive reserve (e.g. attention and perceptual-motor function).
  Arms: Music Intervention
Other: Reading Intervention — After training, caregivers will deliver the reading intervention to the person with dementia whom they care for. The reading intervention will include: a) the caregiver reading aloud to the person they are caring for; b) the person with dementia reading aloud to their caregiver; and c) discussion of the text and personal responses. Strategies to engage the person with dementia and to create opportunities for meaningful dialogue will be provided, as well as guidance on selecting reading material that is accessible to the person's level of cognitive impairment.
  Arms: Reading Intervention

SUMMARY:
This international study evaluates the impact of home-based caregiver-delivered music and reading interventions for people with dementia. The project aims to address the need for improved informal dementia care by training family caregivers to utilise a music or reading intervention with the person they are caring for. The interventions aim to decrease behavioural and psychological symptoms of dementia as well as improve quality of life and well being of both people living with dementia and their caregivers. Participants will be allocated into a music intervention group, a reading intervention group or standard care group. In addition, the researchers will seek to determine the cost-effectiveness of using the music intervention.

DETAILED DESCRIPTION:
This three-arm parallel-group randomised controlled trial will involve 495 couples (cohabiting caregivers and people with dementia) across 5 countries. Caregivers allocated to the music or reading intervention groups will be given three 2-hour training sessions in the allocated intervention. They will be asked to deliver the intervention to the person they are caring for 5x weekly for 3 months. Data will be collected prior to implementing the intervention, during the intervention (via diaries kept by the caregivers), after the last week of implementing the intervention and 3-months after implementing the intervention.

The investigators will explore whether caregiver-delivered music or reading activities improve behavioural and psychological symptoms for people living with dementia. The researchers will also seek to find out the impact on other aspects of both the person with dementia and their caregiver's quality of life and well being. Additionally, costs associated with the care of the person with dementia will be evaluated to determine cost-effectiveness of delivering a music intervention.

ELIGIBILITY:
Inclusion Criteria:

* Dyads (cohabiting) who are close in relationship and where one member has a diagnosis of dementia according to ICD-10 criteria (Alzheimer's Disease [AD], Frontotemporal Dementia, Vascular Dementia [VD], Lewy Body Disease, or mixed dementia) as determined by a clinician experienced in diagnosing dementia. Close in relationship refers to a caregiver who may be a sibling, spouse, adult child, friend, niece or nephew or any person who has a close relationship to the person with dementia, that is, anyone who is not a formal paid caregiver.
* Dyads where the person with dementia has a Neuropsychiatric Inventory-Questionnaire (NPI-Q) Score of ≥6 (from a maximum score of 36)

Exclusion Criteria:

* Dyads where either or both the caregiver or person with dementia have significant hearing impairments that are not resolved through the use of a hearing aid device and limit their capacity to enjoy musical experiences
* There will be no further exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline of behavioural and psychological symptoms of participants with dementia at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Neuropsychiatric Inventory Questionnaire (NPI-Q). Severity scores range from 0-36, where higher scores indicate more severe behavioural and psychological symptoms of dementia. Distress scores range from 0-60, where higher values represent higher levels of distress due to symptoms.

SECONDARY OUTCOMES:
Change from baseline of depression in participants with dementia at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Montgomery Asberg Depression Rating Scale (MADRS). Scale scores range from 0-60, where higher scores indicate more severe depression.
Change from baseline of quality of life of participants with dementia at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Quality of Life - Alzheimer's Disease (QoL-AD) scale. Scale scores range from 13-52, where higher scores indicate higher quality of life.
Change from baseline of depression in caregiver participants at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Patient Health Questionnaire-9 (PHQ-9). Scale scores range from 0-27, where scores greater than 20 indicate severe depression.
Change from baseline of resilience in caregiver participants at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Resilience Scale-14 (RS-14). Scale scores range from 14-98, where higher scores indicate higher resilience.
Change from baseline in caregiver competence of caregiver participants at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Short Sense of Competence Questionnaire (SSCQ). Scale scores range from 7-35, where higher scores indicate higher sense of competence.
Change from baseline in quality of life of caregiver participants at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Assessment of Quality of Life-6D (AQOL-6D).
Change from baseline in quality of the relationship between caregiver and person with dementia at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Quality of Caregiver-Patient Relationship (QCPR). Scale scores range from 14-70, where higher scores indicate a higher quality of relationship.
Change from baseline in quality of adjusted life-years of caregiver and person with dementia at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the EuroQoL Instrument (EQ-5D-5L).
Change from baseline in resource use of both caregiver and person with dementia (cost-effectiveness) at post-intervention and 6-month follow-up | baseline, 12-weeks (primary time-point), and 6-months after intervention commencement (follow-up)
  Measured by the Resource Utilization in Dementia (RUD).

OTHER OUTCOMES:
Intervention dosage throughout intervention | Throughout the 12-weeks caregiver-delivered intervention (at least 5x per week)
  Measured using the tailored diary for caregivers to record the duration of music or reading intervention use, responses of the person with dementia and details of activities used.
Caregivers' experiences of delivering the music and reading interventions | 12-weeks (primary time point)
  Measured using post-intervention qualitative interviews with caregivers to capture descriptions of their experience of delivering the intervention and data to fine-tune the training, research design and the protocol.
Caregivers' experiences and reactions to the music and reading intervention training sessions | Post intervention training sessions at 1-week, 3-weeks, and 6-weeks
  Measured using a short questionnaire.
Caregivers' adherence to programme and ability to apply the learning from the training sessions in their day-to-day caring | Throughout the 12-weeks caregiver-delivered intervention (at least 5x per week)
  Measured using the tailored diary for caregivers to record the duration of music or reading intervention use, responses of the person with dementia and details of activities used
Change from baseline of cognition of participants with dementia at post-intervention to explore relationship between cognitive decline, behavioural and psychological symptoms of dementia, depression and response to different conditions | baseline and 12-weeks (primary time-point, post-intervention)
  Measured using the Mini-Mental State Examination (MMSE). Scores Higher scores indicate better cognitive capacity with scores of 24-30 indicating no cognitive impairment; 19-23 indicating mild cognitive impairment; 10-18 indicating moderate cognitive impairment; and scores <10 indicating severe cognitive impairment.
Adverse events | Phone calls at weeks 2, 4, 6, 8, 10, 12
  Adverse events will be measured throughout the 12-week intervention period for all groups via fortnightly phone calls. Participants will be asked about any adverse events they may have experienced, including hospitalisations, unexpected GP appointments or negative responses to the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Felicity Baker, Professor, Study Director — University of Melbourne
Locations (5):
- The University of Melbourne, Melbourne, Australia
- University of Applied Sciences Würzburg-Schweinfurt, Würzburg, Germany
- Norwegian Academy of Music, Oslo, Norway
- University of Physical Education in Krakow, Krakow, Poland
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the Australian Code for Responsible Conduct of Research (Universities Australia, 2018), all data will be retained for retrieval and re-use in future research where participant permission is granted. Data made available will include individual-level deidentified participant data, reports on adverse events, and deidentified interview transcripts.
Supporting Information: Study Protocol
Time Frame: Following project completion, de-identified anonymised data will be made available (with participant consent). According to the GDPR, the consortium have agreed for reused for 10 years after the project has been completed.
Access Criteria: Data will be made available on the Australian Data Archive https://ada.edu.au and listed on Research Australia's https://researchaustralia.org website to facilitate access for future research.

REFERENCES:
- [Derived] Bukowska AA, Janus E, Soo VP, Smrokowska-Reichmann A, Hsu MH, Stensaeth KA, Odell-Miller H, Tamplin J, Wosch T, Sousa TV, Lamb KE, Braat S, Baker FA. Relationship between dementia diagnostic characteristics and severity of depressive symptoms in a cross-sectional analysis of HOMESIDE baseline data. Sci Rep. 2025 Oct 21;15(1):36643. doi: 10.1038/s41598-025-20385-z. PMID 41120472
- [Derived] Baker FA, Pac Soo V, Bloska J, Blauth L, Bukowska AA, Flynn L, Hsu MH, Janus E, Johansson K, Kvamme T, Lautenschlager N, Miller H, Pool J, Smrokowska-Reichmann A, Stensaeth K, Teggelove K, Warnke S, Wosch T, Odell-Miller H, Lamb K, Braat S, Sousa TV, Tamplin J. Home-based family caregiver-delivered music and reading interventions for people living with dementia (HOMESIDE trial): an international randomised controlled trial. EClinicalMedicine. 2023 Oct 2;65:102224. doi: 10.1016/j.eclinm.2023.102224. eCollection 2023 Nov. PMID 38106552
- [Derived] Pac Soo V, Baker FA, Sousa TV, Odell-Miller H, Stensaeth K, Wosch T, Bukowska AA, Tamplin J, Lautenschlager N, Braat S, Lamb KE. Statistical analysis plan for HOMESIDE: a randomised controlled trial for home-based family caregiver-delivered music and reading interventions for people living with dementia. Trials. 2023 May 8;24(1):316. doi: 10.1186/s13063-023-07327-8. PMID 37226214
- [Derived] Baker FA, Bloska J, Braat S, Bukowska A, Clark I, Hsu MH, Kvamme T, Lautenschlager N, Lee YC, Smrokowska-Reichmann A, Sousa TV, Stensaeth KA, Tamplin J, Wosch T, Odell-Miller H. HOMESIDE: home-based family caregiver-delivered music and reading interventions for people living with dementia: protocol of a randomised controlled trial. BMJ Open. 2019 Nov 19;9(11):e031332. doi: 10.1136/bmjopen-2019-031332. PMID 31748300